CLINICAL TRIAL: NCT02822677
Title: The Distribution of Irritable Bowel Syndrome (IBS) Subtypes, Chinese Medicine Pattern and Host-gut Microbiota Metabolic Interactions Associated With IBS Subtypes
Brief Title: A Cross-sectional Study on IBS Subtypes, Chinese Medicine Pattern and Host-gut Microbiota Metabolic Interactions
Status: Completed | Type: Observational
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Chair Professor, Hong Kong Baptist University
Other Study IDs: HKBUIBS2016
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — Serum: The participants will be instructed to meet fasting for the blood sample collection and 15ml whole blood will be drawn from the participants.
  Stool: Fecal samples should be naturally excreted from subjects (500ml at least) and should be collected without mixing with urine, sanitizer and sewage.
  Urine: Mid-stream morning urine will be collected.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators will conduct a cross-sectional study to discovery the distribution of IBS subtypes who would like to seek TCM treatment and their TCM patterns. At the same time, the investigators will also collect the serum, urine and stool samples of the participants to explore the host-gut microbiota metabolic interactions associated with IBS subtypes.

DETAILED DESCRIPTION:
It is a cross-sectional study to discovery the distribution of IBS subtypes who would like to seek CM treatment and their CM patterns.Serum, urine and stool samples of the participants will be collected from 400-600 IBS participants to explore the host-gut microbiota metabolic interactions associated with IBS subtypes. The primary outcome will be the distribution of IBS subtype and their CM pattern in Hong Kong population. Secondary outcomes will be the host-gut microbiota metabolic interactions associated with IBS subtypes, the relationship between CM pattern and their microbiota and metabolic profiling. The relationship between IBS subtype distribution and other predetermined factors will be assessed, including gender, age, weight, Body Mass Index (BMI), dietary habit, education, economical status, the overall and individual IBS Symptom Severity Scale (IBS-SSS), syndrome of Chinese medicine, QoL assessment and Bristol Stool Scale.For those who had fulfillment of the Structured Clinical Interview for DSM-5 Disorders-(SCID-5), the Hamilton Depression Rating Scale (HAMD-17), Clinical Global Impression-severity (CGI-S), and Self-Rating Depression Scale (SDS) will also be assessed. After the collection of serum, urine and stool samples, bacterial total DNA will be extracted, purified,concentrated,dried and stored for further fecal 16s rRNA sequencing analysis. A number of parameters, including serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphate (ALP) et al., will be measured in serum. Total BA and BA profiles in serum and feces will be tested as well.

ELIGIBILITY:
Inclusion Criteria:

* 1) meet of diagnosis of IBS(ROME 4); 2) age of 18 to 65 years (inclusive); 3) IBS Symptom Severity Scale [17] (IBS-SSS) > 75 points (a range of 0-500 points of VAS on five questions) at baseline and during the 2-week run-in period; 4) Normal colonic evaluation (colonoscopy or barium enema) within 5 years; 5) Written informed consent.

Exclusion Criteria:

* 1) pregnancy or breast-feeding; 2) medical history of inflammatory bowel diseases, carbohydrate malabsorption, hormonal disorder, known allergies to food additives, and/or any other serious diseases; 3) Having suicidal ideas or attempts or aggressive behavior; 4) Use of medications known to influence gastrointestinal transit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBS Patients
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
the Distribution of IBS Subtype and Their CM Pattern in Hong Kong Population. | one year

SECONDARY OUTCOMES:
the Host-gut Microbiota Metabolic Interactions Associated with IBS Subtypes | one year
the Relationship Between CM Pattern and Their Microbiota | one year
the relationship between CM pattern and metabolic profiling | one year

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-xiang Bian, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine, Hong Kong Baptist University, Hong Kong, Hong Kong, China